CLINICAL TRIAL: NCT00559520
Title: The Role of Preoperative Oral Immunonutrition in Major Vascular Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Screening
Other Study IDs: PHRC 2004
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Undernutrition
Keywords: Patients; Suffering; Undernutrition; Requiring; Vascular; Surgery
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Impact (Active Comparator): patient receiving 3 drinks "Impact" a day during 5 days before surgery
  Interventions: Dietary Supplement: Impact
- Oral Impact (Experimental): Patient receiving 3 drinks "Oral Impact" a day during 5 days before surgery
  Interventions: Dietary Supplement: Oral Impact

INTERVENTIONS:
Dietary Supplement: Impact — Patient receiving 3 drinks "Impact" a day during 5 days before surgery
  Arms: Impact
Dietary Supplement: Oral Impact — Patient receiving 3 drinks "Oral Impact" a day during 5 days before surgery
  Arms: Oral Impact

SUMMARY:
The role of preoperative oral immunonutrition in major vascular surgery.

The mean purpose of this study was to determine the prevalence of post-operative infection complications after major vascular surgery in group of patients with preoperative oral immunonutrition.

This group was compared to a control group.

Secondary purpose was to evaluate the effect of preoperative oral immunonutrition on postoperative mortality (30 days), the medium length of stay in the hospital and the cost of treatment in the two groups

ELIGIBILITY:
Inclusion Criteria:

* Intervention planned since at least 5 days before surgery
* Duration of hospitalization of at least 5 days

Exclusion Criteria:

* Pregnant or lactating woman
* Patient with severe renal insufficiency
* Patient under 18 years old
* Patient infected with HIV,hépatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2002-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Weight | before surgery, five days and thirty days after surgery
Arisen of an infectious complication | during the period of 30 days following the surgery
Arisen of non infectious complication | during the period of 30 days following the surgery

SECONDARY OUTCOMES:
Primary and secondary permeability | at 5 and 30 days after surgery
Pain | at 5 and 30 days after surgery
Healing | at 5 and 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michel BATT, Professeur, Principal Investigator — Department of Vascular Surgery, CHU de NICE
Locations (1):
- CHU de NICE, Department of Vascular Surgery, Nice, France

REFERENCES:
- [Background] Gallagher-Allred CR, Voss AC, Finn SC, McCamish MA. Malnutrition and clinical outcomes: the case for medical nutrition therapy. J Am Diet Assoc. 1996 Apr;96(4):361-6, 369; quiz 367-8. doi: 10.1016/s0002-8223(96)00099-5. PMID 8598437
- [Background] Bauer J, Capra S, Ferguson M. Use of the scored Patient-Generated Subjective Global Assessment (PG-SGA) as a nutrition assessment tool in patients with cancer. Eur J Clin Nutr. 2002 Aug;56(8):779-85. doi: 10.1038/sj.ejcn.1601412. PMID 12122555
- [Background] Hill GL, Blackett RL, Pickford I, Burkinshaw L, Young GA, Warren JV, Schorah CJ, Morgan DB. Malnutrition in surgical patients. An unrecognised problem. Lancet. 1977 Mar 26;1(8013):689-92. doi: 10.1016/s0140-6736(77)92127-4. PMID 66485
- [Background] Arora NS, Rochester DF. Respiratory muscle strength and maximal voluntary ventilation in undernourished patients. Am Rev Respir Dis. 1982 Jul;126(1):5-8. doi: 10.1164/arrd.1982.126.1.5. PMID 7091909
- [Background] Heymsfield SB, Bethel RA, Ansley JD, Gibbs DM, Felner JM, Nutter DO. Cardiac abnormalities in cachectic patients before and during nutritional repletion. Am Heart J. 1978 May;95(5):584-94. doi: 10.1016/0002-8703(78)90300-9. No abstract available. PMID 416704
- [Background] Reilly JJ Jr, Hull SF, Albert N, Waller A, Bringardener S. Economic impact of malnutrition: a model system for hospitalized patients. JPEN J Parenter Enteral Nutr. 1988 Jul-Aug;12(4):371-6. doi: 10.1177/0148607188012004371. PMID 3138447
- [Background] Gianotti L, Braga M, Nespoli L, Radaelli G, Beneduce A, Di Carlo V. A randomized controlled trial of preoperative oral supplementation with a specialized diet in patients with gastrointestinal cancer. Gastroenterology. 2002 Jun;122(7):1763-70. doi: 10.1053/gast.2002.33587. PMID 12055582
- [Background] Gianotti L, Braga M, Frei A, Greiner R, Di Carlo V. Health care resources consumed to treat postoperative infections: cost saving by perioperative immunonutrition. Shock. 2000 Sep;14(3):325-30. doi: 10.1097/00024382-200014030-00015. PMID 11028551
- [Background] Robinson G, Goldstein M, Levine GM. Impact of nutritional status on DRG length of stay. JPEN J Parenter Enteral Nutr. 1987 Jan-Feb;11(1):49-51. doi: 10.1177/014860718701100149. PMID 3102782
- [Background] Chima CS, Barco K, Dewitt ML, Maeda M, Teran JC, Mullen KD. Relationship of nutritional status to length of stay, hospital costs, and discharge status of patients hospitalized in the medicine service. J Am Diet Assoc. 1997 Sep;97(9):975-8; quiz 979-80. doi: 10.1016/S0002-8223(97)00235-6. PMID 9284874
- [Background] Braunschweig C, Gomez S, Sheean PM. Impact of declines in nutritional status on outcomes in adult patients hospitalized for more than 7 days. J Am Diet Assoc. 2000 Nov;100(11):1316-22; quiz 1323-4. doi: 10.1016/S0002-8223(00)00373-4. PMID 11103653
- [Background] Lewis SJ, Egger M, Sylvester PA, Thomas S. Early enteral feeding versus "nil by mouth" after gastrointestinal surgery: systematic review and meta-analysis of controlled trials. BMJ. 2001 Oct 6;323(7316):773-6. doi: 10.1136/bmj.323.7316.773. PMID 11588077
- [Background] Spark JI, Robinson JM, Gallavin L, Gough MJ, Homer-Vanniasinkam S, Kester RC, Scott DJ. Patients with chronic critical limb ischaemia have reduced total antioxidant capacity and impaired nutritional status. Eur J Vasc Endovasc Surg. 2002 Dec;24(6):535-9. doi: 10.1053/ejvs.2002.1755. PMID 12443751
- [Background] Evoy D, Lieberman MD, Fahey TJ 3rd, Daly JM. Immunonutrition: the role of arginine. Nutrition. 1998 Jul-Aug;14(7-8):611-7. doi: 10.1016/s0899-9007(98)00005-7. PMID 9684265
- [Background] Kirk SJ, Barbul A. Role of arginine in trauma, sepsis, and immunity. JPEN J Parenter Enteral Nutr. 1990 Sep-Oct;14(5 Suppl):226S-229S. doi: 10.1177/014860719001400514. No abstract available. PMID 2232107
- [Background] Wu D, Meydani SN. n-3 polyunsaturated fatty acids and immune function. Proc Nutr Soc. 1998 Nov;57(4):503-9. doi: 10.1079/pns19980074. PMID 10096109
- [Background] Beale RJ, Bryg DJ, Bihari DJ. Immunonutrition in the critically ill: a systematic review of clinical outcome. Crit Care Med. 1999 Dec;27(12):2799-805. doi: 10.1097/00003246-199912000-00032. PMID 10628629
- [Background] Heyland DK, Novak F, Drover JW, Jain M, Su X, Suchner U. Should immunonutrition become routine in critically ill patients? A systematic review of the evidence. JAMA. 2001 Aug 22-29;286(8):944-53. doi: 10.1001/jama.286.8.944. PMID 11509059
- [Background] Heys SD, Walker LG, Smith I, Eremin O. Enteral nutritional supplementation with key nutrients in patients with critical illness and cancer: a meta-analysis of randomized controlled clinical trials. Ann Surg. 1999 Apr;229(4):467-77. doi: 10.1097/00000658-199904000-00004. PMID 10203078
- [Background] Bower RH, Cerra FB, Bershadsky B, Licari JJ, Hoyt DB, Jensen GL, Van Buren CT, Rothkopf MM, Daly JM, Adelsberg BR. Early enteral administration of a formula (Impact) supplemented with arginine, nucleotides, and fish oil in intensive care unit patients: results of a multicenter, prospective, randomized, clinical trial. Crit Care Med. 1995 Mar;23(3):436-49. doi: 10.1097/00003246-199503000-00006. PMID 7874893
- [Background] Tepaske R, Velthuis H, Oudemans-van Straaten HM, Heisterkamp SH, van Deventer SJ, Ince C, Eysman L, Kesecioglu J. Effect of preoperative oral immune-enhancing nutritional supplement on patients at high risk of infection after cardiac surgery: a randomised placebo-controlled trial. Lancet. 2001 Sep 1;358(9283):696-701. doi: 10.1016/s0140-6736(01)05836-6. PMID 11551575
- [Background] Melchior JC. [How to assess preoperative nutritional status?]. Ann Fr Anesth Reanim. 1995;14 Suppl 2:19-26. doi: 10.1016/s0750-7658(95)80098-0. French. PMID 7486330
- [Background] Johnson JA, Cogbill TH, Strutt PJ, Gundersen AL. Wound complications after infrainguinal bypass. Classification, predisposing factors, and management. Arch Surg. 1988 Jul;123(7):859-62. doi: 10.1001/archsurg.1988.01400310073012. PMID 3382352